CLINICAL TRIAL: NCT03198598
Title: Effects of Yoga Practice in Multiple Sclerosis Patients: a Multidimensional Approach
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HIAE_EscleroseMultipla_Yoga
Record Dates: First submitted 2017-04-04; First posted 2017-06-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MS patients with EDSS from 0 to 5.5 for yoga (Experimental): Three months of Iyengar Yoga practice.
  Interventions: Behavioral: Iyengar Yoga
- MS patients with EDSS from 0 to 5.5 for control (No Intervention)
- MS patients with EDSS from 6 to 8 for yoga (Experimental): Receive a smartphone application that has an eight-week program including meditation practices, Yoga exercises that can be done in a seated or laid position and daily care tips
  Interventions: Behavioral: Yoga app
- MS patients with EDSS from 6 to 8 for control (No Intervention)
- Healthy subjects (No Intervention)

INTERVENTIONS:
Behavioral: Iyengar Yoga — The patients are going to practice Yoga two times per week during 60 minutes each composed by: 40 minutes of postures, 10 minutes of breathing exercises and 10 minutes of meditation. The proposed Yoga postures will depend on disease severity and will be adapted according to each patient.
  Arms: MS patients with EDSS from 0 to 5.5 for yoga
Behavioral: Yoga app — The patients showing EDSS scores above 6.0 will be divided in two groups of 20. Due to their movements limitations it is not possible to perform a regular Yoga class. In this case they will receive a smartphone application that has an eight-week program including meditation practices, Yoga exercises that can be done in a seated or laid position and daily care tips.
  Arms: MS patients with EDSS from 6 to 8 for yoga

SUMMARY:
In this study the investigators will evaluate the effects of yoga practice on multiple sclerosis patients and healthy controls for fatigue, quality of life, movement, cognition, brain activity, self-efficacy, stress, anxiety, depression, affective states and immunological response. To investigate the effects of yoga training delivered by a yoga instructor or through a smartphone application, the investigators will use a multidimensional approach that comprises of: evaluation of neuropsychological, quality of life and affective aspects, structural and functional magnetic resonance imaging, functional near infrared spectroscopy (fNIRS) combined with movement analysis (gait, strength, balance etc.) and analysis of the immune response.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is one of the most common neurological diseases, which is a cause of disability in young adults. Approximately 60% of the patients will not be able to walk at some point in the disease course. This brings important implications for patients' and family members' quality of life and financial cost to the society. In spite of the clinical significance of MS, its pathophysiology is not completely understood. Many researches have been investigating the role of B and T lymphocytes, the extension of central nervous system lesions and brain activation through neuroimage, separately. A multidimensional approach is necessary for the understanding of MS mechanisms and to verify the effects of therapies, including non-conventional ones, such as yoga. Yoga has been reported as a safe and low coast practice which may be more accessible to MS patients than other types of exercises. In patients with MS there are few well controlled studies, which indicate for example, improvements in fatigue, mobility, gait and humor.

Objectives: To evaluate the effects of yoga practice in MS patients with different EDSS (Expanded Disability Status Scale) scores and healthy controls in aspects such as fatigue, quality of life, movement, cognition, brain activity, self-efficacy, stress, anxiety, depression, affective states and immune response through the analysis of cytokines and B lymphocytes antibody production.

Method: the investigators will apply a multidimensional approach which involves neuropsychological, quality of life and affective aspects evaluation, structural and functional magnetic resonance imaging, near infrared spectroscopy (NIRS) combined with movement analysis (gait, strength, balance etc.), measurements of cytokines and B cells antibody production, comparing MS patients with different scores in the EDSS and healthy controls before and after receiving yoga training delivered by a yoga instructor or through a smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis patients from 18 to 60 years of age, currently in stable immunomodulatory or immunosuppression therapy with no signs of clinical or radiological disease activity for the last 6 months.
* EDSS from 0 to 8

Exclusion Criteria:

* presents clinical or radiological disease activity for the last 6 months
* no cognitive capacity to understand the written informed consent form

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2026-12-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Improvement of overall MS impact in patients life | 3 months
  Multiple Sclerosis Impact Scale-29 (MSIS-29 - Hobart J et al, 2001);
Cognition in MS | 3 months
  Brief International Cognitive Assessment for MS with will evaluate executive function in MS patients
Fatigue in MS | 3 months
  Modified Fatigue Impact Scale (MFIS - Pavan et al., 2007)- evaluates the level of fatigue in everyday life.
Self-efficacy in MS | 3 months
  MS Self-Efficacy Scale (MSSE - Schwartz et al., 1996)- to evaluate self-efficacy in everyday life

SECONDARY OUTCOMES:
Cyytokine levels | 3 months
  The immune system response to the intervention will be evaluated through cytokines levels
Correlation between gait and hemodynamic response | 3 months
  The participants will be asked to perform a dual-task inside the gait lab. During the task, we will acquire hemoynamic response from dorso-lateral, SMA, pre-motor and motor cortex using functional near infrared spectroscopy technology (fNIRS). The gait parameters (e.g: step length, joint angles and velocity) recorded will be correlated with the cortical activations taken from the fNIRS.
Motor agility | 3 months
  9-hole Peg Test (9-HPT - Grice et al., 2003);
Awareness and attention | 3 months
  Mindful attention awareness scale (Brown & Ryan 2003);
Lymphocyte B activity | 3 months
  The immune system response to the intervention will be also evaluated through the Lymphocyte B activity
Walking speed | 3 months
  Timed 25 foot walk - (National Multiple Sclerosis Society, 2016);
Ability to stand up and walk | 3 month3
  Timed up & go (Podsiadlo & Richardson, 1991);
Hands strenght | 3 months
  Hand grip (Godoy, 2005 );
Self-compassion | 3 months
  Self-compassion scale (Neff, 2003);
Affects | 3 months
  Positive and Negative Affect Schedule (PANAS - Carvalho, 2013);

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No